CLINICAL TRIAL: NCT03316287
Title: EVidenced Based Management of Hearing Impairments: Public Health pΟlicy Making Based on Fusing Big Data Analytics and simulaTION
Brief Title: Big Data Supporting Public Health Hearing Policies
Acronym: EVOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17/0064
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids; Calibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hearing aid + mobile phone (Experimental)
  Interventions: Device: Hearing aid; Device: Mobile phone
- Hearing aid + mobile phone + biosensor (Experimental)
  Interventions: Device: Hearing aid; Device: Mobile phone; Device: Sensor

INTERVENTIONS:
Device: Hearing aid — Smart hearing aid to allow collection of real time hearing aid usage data
Device: Mobile phone — Mobile phone linked with the hearing aids to allow users to change the device settings and perform additional listening tests
Device: Sensor — Wearable biosensor for the collection of physiological data
  Arms: Hearing aid + mobile phone + biosensor

SUMMARY:
Hearing Loss (HL) affects over 5% of the world's population (WHO 2014) and is the 5th leading cause of Years Lived with Disability. HL is currently managed with Hearing Aids (HAs), i.e. programmable sound amplification devices that are worn by the hearing impaired subjects to address their hearing difficulties. HA use however is often problematic, costly and with poor overall benefits. The holistic management of HL requires appropriate public health policies for HL prevention, early diagnosis, long-term treatment and rehabilitation; detection and prevention of cognitive decline; and socioeconomic inclusion of HL patients. Currently the evidential basis for forming such policies is limited.

The EVOTION project proposes to address this by collecting and analysing a big set of heterogeneous data, including HA usage, audiological, physiological, cognitive, clinical and medication, personal, behavioural, life style, occupational and environmental data.

This will be done by:

i. accessing big datasets of existing HA user data from the EVOTION clinical partners (UCL/UCLH and GST in the UK; OTICON in Denmark) ii. collection of prospective HA user data who will be recruited to the prospective EVOTION study and who will undergo some additional assessments iii. collection of real time dynamic data of the human participant HA users who will be given a smart phone with different apps (auditory tests; auditory training), sensors (recording of heart rate, blood pressure, respiratory rate etc.) and smart HAs (recording environmental factors such as noise levels, type of noise etc.) so that real life contextual factors that affect HA usage and outcome can be identified.

These data will be analysed with big data analysis/data mining techniques in order to identify relationships between these in order to use this information to derive and support public health decisions.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Basic understanding of oral and written English
* Unilateral and/or bilateral mild to severe sensorineural hearing loss
* Willing to use smart hearing aids for at least 2 hours daily on average
* Willing/capable to use a mobile phone

Exclusion Criteria:

* Dementia (MoCA<22 )
* Not agreeing or able to attend for f/u appointments
* Not agreeing or able to use HA >2 hours daily (average)
* Not sufficient vision to use smartphone ap

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1080 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in "Glasgow Hearing Aid Benefit Profile" at 8 weeks | Baseline (i.e. before the patient receives a hearing-aid) and at 8 weeks after receiving a hearing-aid

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St. Thomas' Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Dritsakis G, Kikidis D, Koloutsou N, Murdin L, Bibas A, Ploumidou K, Laplante-Levesque A, Pontoppidan NH, Bamiou DE. Clinical validation of a public health policy-making platform for hearing loss (EVOTION): protocol for a big data study. BMJ Open. 2018 Feb 15;8(2):e020978. doi: 10.1136/bmjopen-2017-020978. PMID 29449298